CLINICAL TRIAL: NCT04427579
Title: Anxiety and Depression in COPD; Prevalence, Detection and Prognosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Akershus (Other)
Collaborators: University of Oslo (Other); LHL Hospital Gardermoen (Unknown); Priory Hospital Altrincham (Unknown)
Responsible Party: Principal Investigator, Gunnar Einvik, Post-doc candidate, MD, University Hospital, Akershus
Other Study IDs: 2018/149
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: COPD; Anxiety Disorders; Depressive Disorder
Keywords: Metacognitions; Hospital Anxiety and Depression Scale
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Anxiety Disorders; Depressive Disorder; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The current cohort study of 300 stable COPD patients aims to assess the following topics:

* The prevalence of anxiety and depressive disorders in patients with COPD
* The screening properties of Hospital Anxiety and Depression Scale in patients with COPD
* The prognostic influence by anxiety or depressive symptoms and anxiety or depressive disorder.
* whether characterization of 1) affective aspects of dyspnea symptoms or 2) persistent styles of thinking (worry or rumination) and metacognitions that drive these may improve the current recommendation of screening for anxiety and depression in COPD in relation to its clinical relevance on functional status and three year outcome

ELIGIBILITY:
Inclusion Criteria:

* Participant in in-hospital pulmonary rehabilitation at LHL-hospital Gardermoen
* Diagnosis of COPD

Exclusion Criteria:

* Acute exacerbated phase of COPD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults referred to and initiating a 2-4 weeks in-hospital rehabilitation course.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
COPD exacerbation rate | 3 years
  The number of moderate or severe exacerbations
Mortality rate | 3 years
  The number of deaths

SECONDARY OUTCOMES:
Assessment of Health-related Quality of Life With RAND-36 | 3 years
  The total score and subscale scores on RAND 36

OTHER OUTCOMES:
The prevalence of anxiety disorder | 1 year
  Clinically diagnosed anxiety disorders
The prevalence of depressive disorder | 1 year
  Clinically diagnosed depressive disorder

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Einvik, PhD, Principal Investigator — University Hospital, Akershus
Locations (1):
- LHL-hospital Gardermoen, Jessheim, Norway

IPD SHARING:
Plan to Share IPD: No